CLINICAL TRIAL: NCT07316478
Title: RCT of Stress Management and Mindfulness Intervention for Patients With Sickle Cell Disease
Brief Title: Stress Management and Mindfulness Intervention for Patients With Sickle Cell Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Melissa Hunt, PhD, Associate Director of Clinical Training, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 859513
Record Dates: First submitted 2025-12-02; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; SCD; Mindfulness; Behavioral Health; stress management; cognitive behavioral therapy; deep diaphragmatic breathing; relaxation training
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hemoglobin, Sickle

STUDY DESIGN:
Intervention Model Description: Waitlist control followed by crossover to active treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): 6 week intervention focused on: How psychological stress affects health and SCD pain crises Deep diaphragmatic breathing and basic relaxation skills to lower stress and improve pain management CBT techniques to rethink situations, reduce stress, and respond less reactively Practice identifying unhelpful thoughts and replacing them with more balanced ones Self-Care & Barriers to Change Learn ways to build more wellness activities into daily life.
  Navigating the ER & Medical Encounters. Learn effective ways to communicate with doctors and nurses unfamiliar with SCD Mindfulness Meditation
  Interventions: Behavioral: Stress Management and Mindfulness Intervention for Patients with Sickle Cell Disease
- Waitlist Control (No Intervention): Participants in the waitlist control will receive no treatment for 6 weeks. After completing the follow-up measures, they will be crossed over to active treatment.

INTERVENTIONS:
Behavioral: Stress Management and Mindfulness Intervention for Patients with Sickle Cell Disease — This is a behavioral health intervention drawing from Cognitive Behavioral Therapy, Mindfulness Techniques, Relaxation Training and Assertiveness training.
  Arms: Immediate Treatment

SUMMARY:
The purpose of this research is to determine whether a new stress management and mindfulness program can improve quality of life in individuals with sickle cell disease. The program is based on a number of empirically supported treatments including techniques from cognitive-behavioral therapy like overcoming motivational barriers to self-care, learning to see things as accurately as possible, practicing assertive communication, relaxation exercises like deep slow breathing, mindfulness meditation, and other stress management strategies.

DETAILED DESCRIPTION:
After consenting and completing the baseline measures, participants will be assigned (like flipping a coin) to the immediate treatment group or the control group. The immediate treatment group will participate in the intervention for six weeks while the control group waits. At the end of six weeks, both groups will complete the measures again, and then the control group will have a chance to participate in the intervention. See table below for the timeline of the study for each group.

Study Stage Immediate Intervention Group Waitlist Control Group

1. Baseline Measures - Complete online demographic, mood, and symptom questionnaires

   * May skip any questions
   * Study team emails to confirm participation Same as Immediate Group
2. Randomization (like flipping a coin) Receive email stating you were assigned to the Immediate Group and will begin the program right away Receive email stating you were assigned to the Waitlist Group and will begin the program after 6 weeks Weeks 1-6 Attend six weekly 1-hour group sessions (in person on the campus of the University of Pennsylvania in room 450 of the NBS building located at 425 S. University Avenue or via Zoom) Waiting period (no sessions yet) End of Week 6 Complete symptom measures again and provide feedback on the program Complete symptom measures at the end of the waiting period Weeks 7-12 No additional sessions during this time Attend six weekly 1-hour group sessions (in person in NBS 450 or via Zoom) End of Week 12 - Complete symptom measures again and provide feedback on the program Final Follow-Up (3 months after completing the program) Complete the symptom questionnaires one last time Complete the symptom questionnaires one last time

Intervention: The intervention is a stress management and mindfulness-based program developed and led by Dr. Melissa Hunt, who is a licensed clinical psychologist with expertise in chronic health conditions and mindfulness interventions. She will be assisted by four research coordinators who are undergraduate psychology majors at the University of Pennsylvania. Participants will also have access to an app called Blackfulness. It is a mindfulness meditation app designed specifically for black people. The in person sessions will take place in person at The Neural and Behavioral Sciences (NBS) Building (425 S University Ave, Philadelphia, PA 19104) Room 450. Remote sessions will take place virtually via Zoom video conferencing. People who elect the in person sessions may choose to attend some sessions remotely if weather or health necessitates it.

Week Focus Goals

1 Stress, Health, and Pain Education • Learn how psychological stress affects health and SCD pain crises

* Learn deep diaphragmatic breathing and basic relaxation skills to lower stress and improve pain management 2 Cognitive Therapy Skills • Learn CBT techniques to rethink situations, reduce stress, and respond less reactively
* Practice identifying unhelpful thoughts and replacing them with more balanced ones 3 Self-Care & Barriers to Change • Explore self-care strategies (sleep, exercise, wellness habits)
* Discuss barriers to self-care and ambivalence about change
* Learn ways to build more wellness activities into daily life. 4 Navigating the ER & Medical Encounters • Learn effective ways to communicate with doctors and nurses unfamiliar with SCD
* Review suggested scripts and role-play interactions with medical personnel
* Practice advocacy skills to make sure your voice is heard 5 Mindfulness Meditation I • Introduction to mindfulness practices that decrease emotional and physical reactivity
* Build self-compassion skills
* Optional use of the Blackfulness app for between-session practice (requires agreeing to the app's privacy policies) 6 Mindfulness Meditation II & Mindful Movement • Continue mindfulness practice, including gentle mindful movement and stretching
* Learn ways to integrate mindfulness into daily routines

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Diagnosed with sickle cell disease.
* Live within 90 minutes of Philadelphia

Exclusion Criteria:

- Severe depression or suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
PROMIS-57 | Baseline, 6 weeks, 3 month follow-up
  PROMIS-57 Profile (PROMIS Health Organization, 2020) offers a broad assessment of health-related quality of life (HRQoL) across multiple domains such as physical function, anxiety, depression, fatigue, and sleep disturbance
ASCQ-Me | Baseline, 6 weeks and 3 month follow-up
  Quality of life in adults with SCD is comprehensively measured by the ASCQ-Me tool (ASCQ-Me User's Manual, American Institutes for Research, 2017), covering emotional distress, pain impact, and sleep disturbances, and validated for use in both clinical and research settings. We will be using the Pain Impact Scale (ASCQ-Me v2.0 Pain Impact - American Institutes for Research, 2017) which assesses how much pain limits daily activities and overall function.

SECONDARY OUTCOMES:
Beck Depression Inventory | Baseline, 6 weeks and 3 month follow-up
  Standard multiple choice measure of depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Melissa G Hunt, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No
To reduce risk of breach of confidentiality